CLINICAL TRIAL: NCT05735886
Title: Impact of Urolithin A Supplementation on Mitochondrial Health of Immune Cells (MitoImmune): a Randomized Trial
Brief Title: Urolithin A Supplementation to Boost Immune Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Goethe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 22.03.AMZ
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: Immune system; mitochondria
MeSH Terms: interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Softgel containing placebo
- Urolithin A (Mitopure) (Active Comparator)
  Interventions: Dietary Supplement: Softgel containing 250mg of Urolithin A (Mitopure)

INTERVENTIONS:
Dietary Supplement: Softgel containing placebo — Single oral dose administration (4 softgels) to be orally administered daily according to the randomization for 28 days
  Arms: Placebo
Dietary Supplement: Softgel containing 250mg of Urolithin A (Mitopure) — Single oral dose administration (4 softgels) to be orally administered daily according to the randomization for 28 days
  Arms: Urolithin A (Mitopure)

SUMMARY:
To show that a natural mitophagy activator (Urolithin A) given orally can modulate mitochondrial activity in immune cells in healthy adults and this results in better immune function

ELIGIBILITY:
Inclusion Criteria:

Healthy Adults that do not suffer from an uncontrolled chronic medical condition that carries metabolic consequences (as assessed by the study physician)

* BMI<35kg/m2
* Provide informed consent
* Adults aged 45-70 years, both genders
* Subjects who have not received any systemic immunosuppression in the past 6 months
* Subjects with any medical condition that in the opinion of the investigators would compromise the study outcome or the safety of the research participant

Exclusion Criteria:

Subject has any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements;

* Clinically significant abnormal laboratory results at screening
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to study ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
* Current gastrointestinal condition which could interfere with the study (e.g. IBS/IBD, diarrhea, acid reflux disease, dysphagia etc.);
* Excessive alcohol consumption and/or a smoker
* Concomitant use of statins
* Engage in regular moderate or vigorous physically activities (i.e. Category 3 as per the IPAQ activity classification)
* Concomitant use of corticosteroids, antibiotics, any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs), immune-boosting(Vitamin C, Zinc) or mitochondrial (COQ10, NAD+) supplements within 45 days prior to screening

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in percentages of CD3+ T-cell immune cell population | 28 days
  In particular, number of CD8+ T memory stem cells (identified by expression of CD8+CD45RA+CCR7+CD95+) and naïve-like T cells (CD8+CD45RA+CCR7+CD95-)
Change in Mitochondrial activity in CD3+ T-cells | 28 days
  Mitochondrial function evaluated as OXPHOS activity via ELISA /Seahorse

SECONDARY OUTCOMES:
Change in pro and anti-inflammatory cytokine levels (IL-6, TNF-a, IL1-B, IL-10) in plasma and/or ex-vivo antigenic stimulation | 28 days
Change in percentages of other immune cell populations (B cells, NK cells, Macrophages, DCs etc.) via flow cytometry | 28 days
Change in Mitochondrial content on CD3 T-cell populations via Mitotracker staining using flow cytometry | 28 days
Change in gene-expression: single cell analysis of CD3+ T-cells | 28 days
Change in PBMC's immune function assessment (mixed-leukocyte reaction (MLR) via antigenic stimulation | 28 days
Change in Lipid profile | 28 days
Epigenetic age of PBMCs (DNA Methylation-derived epigenetic age) | 28 days
Number of adverse events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dominic Denk, MD, Principal Investigator — Universitätsklinikum Frankfurt Medizinische Klinik I
Locations (1):
- Universitätsklinikum Frankfurt, Medizinische Klinik I, Gastroenterologie/Hepatologie; Frankfurt, Germany, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denk D, Singh A, Kasler HG, D'Amico D, Rey J, Alcober-Boquet L, Gorol JM, Steup C, Tiwari R, Kwok R, Arguello RJ, Faitg J, Sprinzl K, Zeuzem S, Nekljudova V, Loibl S, Verdin E, Rinsch C, Greten FR. Effect of the mitophagy inducer urolithin A on age-related immune decline: a randomized, placebo-controlled trial. Nat Aging. 2025 Nov;5(11):2309-2322. doi: 10.1038/s43587-025-00996-x. Epub 2025 Oct 31. PMID 41174221